CLINICAL TRIAL: NCT05449483
Title: A Prospective, Single-center, Single-arm Phase II Clinical Study of the Safety and Efficacy of Tislelizumab Combined With Chemotherapy in the Treatment of Unresectable Esophageal Squamous Cell Carcinoma
Brief Title: Conversion of Tislelizumab Combined With Chemotherapy in Unresectable Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20220333A
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Esophageal Squamous Cell Carcinoma by AJCC V8 Stage; Unresectable
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tislelizumab+ Paclitaxel+Cisplatin (Experimental): Paclitaxel 135mg/m2 , D1; Cisplatin 80mg/m2, D1; tislelizumab 200mg D2 ; totally 2-4 cycles
  Interventions: Drug: tislelizumab+ Paclitaxel + Cisplatin

INTERVENTIONS:
Drug: tislelizumab+ Paclitaxel + Cisplatin — tislelizumab combined with chemotherapy
  Other Names: conversion therapy

SUMMARY:
Whether the introduction of immunotherapy can transform unresectable esophageal cancer into resectable, or even achieve R0 surgical resection, has not been reported yet. We plan to conduct a prospective, single-center, single-arm phase II clinical study of the safety and efficacy of tislelizumab combined with chemotherapy in the treatment of unresectable esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
For patients not eligible for R0 resection (defined as locally advanced unresectable esophageal cancer), preoperative treatment can theoretically transform the tumor into a resectable state. The current significance of transformation therapy is to reduce tumor volume and stage to achieve radical resection, eliminate micrometastases, and prevent a postoperative recurrence. There are few studies on the transformation therapy of esophageal squamous cell carcinoma. We plan to conduct a prospective, single-center, single-arm phase II clinical study of the safety and efficacy of tislelizumab combined with chemotherapy in the treatment of T4a/N3 esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed esophageal squamous cell carcinoma;
2. Unresectable cT4a/N3(stage ⅣA) (AJCC 8 TNM classification);
3. Have a performance status of 0 or 1 on the ECOG Performance Scale;
4. Age 18-75 years old, both men and women;
5. Be willing and able to provide written informed consent/assent for the trial;
6. Demonstrate adequate organ function, all screening labs should be performed within 10 days of treatment initiation;
7. Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours before receiving the study medication's first dose. If the urine test is positive or cannot be confirmed as unfavorable, a serum pregnancy test will be required;
8. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion through repeated biopsies. Newly acquired is defined as a specimen obtained up to 4 weeks (28 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.

Exclusion Criteria:

1. Prior therapy (operation, radiotherapy, immunotherapy, or chemotherapy) for esophageal cancer;
2. Ineligibility or contraindication for esophagectomy;
3. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug;
4. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with the use of disease-modifying agents, corticosteroids, or immunosuppressive drugs);
5. Has severe hypersensitivity and adverse events (≥Grade 3) to any PD-1/PD-L1 inhibitors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
R0 Surgical Resection Rate . | 1 year
  R0 resection rate

SECONDARY OUTCOMES:
Evaluate the rate of pathologic complete response (pCR) to the study regimen | 1 year
  The percentage of pathologic complete response at resection for patients who has completed the study regimen
Evaluate the rate of main pathologic response (MPR) to the study regimen. | 1 year
  Viable tumor comprised ≤ 10% of resected tumor specimens
Objective response rate (ORR) | 1 year
  Partial response is defined as a decrease by 30% or more in sums of longest diameter of measurable target lesions
Disease-free survival (DFS) | 3 years
  DFS is defined as the time interval between the date of enrollment and the date of the first documented evidence of relapse after radical resection at any site or death related to cancer
Overall survival (OS) | 3 years
  Time from the enrollment to death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Hongjing Jiang, MD，phD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Hongjing Jiang, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No